CLINICAL TRIAL: NCT01548677
Title: TRastuzumab in HER2-negative Early Breast Cancer as Adjuvant Treatment for Circulating Tumor Cells (CTC) ("TREAT CTC" Trial)
Brief Title: Efficacy Study of Herceptin to Treat HER2-negative CTC Breast Cancer
Acronym: TREAT-CTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Hoffmann-La Roche (Industry); Janssen Diagnostics, LLC (Industry); SUCCESS (Unknown); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-90091-10093; 2009-017485-23 (EudraCT Number)
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Circulating Tumor Cells
Keywords: Circulating Tumour Cells; HER2 negative primary breast cancer; HER2 positive CTC; Trastuzumab
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- observation (No Intervention): 18 weeks
- Herceptin (trastuzumab) (Experimental): 18 weeks
  Interventions: Drug: trastuzumab

INTERVENTIONS:
Drug: trastuzumab — 8 mg/kg of loading dose IV over 90 minutes for the first cycle, followed by 6 mg/kg IV over 60 minutes every 3 weeks for the 5 subsequent cycles.
  Other Names: endocrine therapy; anti HER2 therapy
  Arms: Herceptin (trastuzumab)

SUMMARY:
This is a randomized phase II trial for patients with HER2 negative primary Breast Cancer (BC) who after completing (neo) adjuvant chemotherapy and surgery have detectable circulating tumour cells (CTC) in peripheral blood.

Eligible patients will be randomised in 1:1 ratio to either the trastuzumab arm or the observation arm.

DETAILED DESCRIPTION:
This is a randomized phase II trial for patients with HER2 negative primary BC who after completing (neo) adjuvant chemotherapy and surgery have detectable CTC(s) in peripheral blood (see eligibility criteria for details). Eligible patients will be randomized in 1:1 ratio to either the trastuzumab arm or the observation arm. Patients randomized to the trastuzumab arm will receive a total of 6 intravenous (IV) administrations every 3 weeks (loading dose 8 mg/kg IV and 5 cycles at 6 mg/kg every 3 weeks). Patients randomized to observation arm shall be observed for 18 weeks. Left ventricular ejection fraction (LVEF) assessment (MUGA and/or ECHO) will be done at baseline for all patients to be randomized. The next LVEF assessments of weeks 9 and week 18 will be done only in patients randomized to trastuzumab arm. Patient registered but with CTC negative result will not be followed-up.

ELIGIBILITY:
* Age ≥ 18 years
* Written informed consent must be given according to ICH/GCP, and national/local regulations
* Availability of peripheral blood draw for CTC blood test
* Tumor block or minimum 10 unstained slides of 4 μm of primary tumor must be available prior to registration for centralized HER2 testing
* ER status available
* Adequately excised non-metastatic and non-relapsed operable primary invasive HER2-negative adeno-carcinoma of the breast *:
* the patient should have completed either
* adjuvant chemotherapy or
* neoadjuvant chemotherapy; in this case residual invasive disease in breast or lymph nodes is required (no complete pathological response) no further adjuvant chemotherapy treatment planned. Prior chemotherapy with doxorubicin restricted to a total dose of 360 mg/m2 or with epirubicin restricted to a total dose of 720 mg/m2 is allowed
* No prior use of anti-HER2 therapy for any reason or immunotherapy for BC
* No concomitant use of bisphosphonate therapy or denosumab for any reason. Prior use of these agents is allowed provided that last treatment has been received at least 4 weeks before registration in the study
* No prior mediastinal irradiation except internal mammary node irradiation for the present BC
* Concomitant adjuvant hormonal therapy or radiotherapy (if applicable) is allowed upon physician's choice
* The interval between definitive surgery (neoadjuvant population) or end of adjuvant chemotherapy (adjuvant population) and registration must be at least 3 weeks but no more than 24 weeks
* No evidence of unresolved or unstable toxicity from prior surgery, adjuvant chemotherapy or radiotherapy
* No history of prior invasive breast carcinoma, except for the BC diagnosed and treated before entry. Unifocal or multifocal unilateral (one breast) or unifocal or multifocal synchronous bilateral breast (both breasts) cancer are acceptable if all invasive tumor foci are HER2- negative. History of previous ductal carcinoma in situ is allowed
* No history of any malignant neoplasms in the past 5 years except for curatively treated basal and squamous cell carcinoma of the skin
* No prior autologous or allogeneic stem cell transplantation
* No history of serious cardiac illness or medical conditions, including but not confined to:
* History of documented congestive heart failure
* High risk uncontrolled arrhythmias
* Angina pectoris requiring anti-anginal medication
* Clinically significant valvular heart disease
* Evidence of transmural infarction on ECG
* Poorly controlled hypertension (e.g. systolic > 180 mm Hg or diastolic > 100 mm Hg)
* No history of other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration
* WHO performance status 0-1
* No concurrent participation in another trial
* No clinically significant active infections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1317 (Actual)
Dates: Start 2013-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
CTC detection | 18 weeks post randomisation
  To compare circulating tumour cell (CTC)detection rate at week 18 between trastuzumab treatment arm and observational arm.

SECONDARY OUTCOMES:
RFI (recurrence free interval) | 2 years after LPI (last patient in)
  Recurrence Free Interval (RFI) (key secondary endpoint) between trastuzumab and observation
IDFS (Invasive Disease Free Survival) | 2 years after LPI
  Invasive Disease Free Survival between trastuzumab and observation
DFS (disease free survival) | 2 years after LPI
  Disease Free survival between trastuzumab and observation
OS (overall survival) | 2 years after LPI
  Overall Survival between trastuzumab and observation
CTC essay | 2 years after LPI
  To evaluate in a clinical trial setting the feasibility, reliability, within patient reproducibility and variability of the assay for CTC(s)
CTC correlation | 2 years after LPI
  To correlate CTC detection rate at baseline and/or week 18 with RFI, IDFS, DFS, OS
safety (cardiac) | 2 years after LPI
  To assess safety, especially cardiac safety, of trastuzumab in women with HER2 negative primary tumors and CTC

CONTACTS AND LOCATIONS:
Overall Officials: Michail Ignatiadis, MD, Principal Investigator — Institut Jules Bordet, Brussels, Belgium; Martine Piccart, MD, Study Chair — Institut Jules Bordet, Brussels, Belgium; Christos Sotiriou, MD, Study Chair — Institut Jules Bordet, Brussels, Belgium; Jean-Yves Pierga, MD, Study Chair — Institut Curie, Paris, France; Brigitte Rack, MD, Study Chair — Ludwig-Maximilians-Universitaet Muenchen - Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe - Innenstadt, Munich, Germany
Locations (80):
- Belgium (9):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Hopital Universitaire Brugmann, Brussels
  - Hopitaux Universitaires Bordet-Erasme - Hopital Universitaire Erasme, Brussels
  - Hôpitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Hopital De Jolimont, Haine-Saint-Paul
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - C.H.U. Sart-Tilman, Liège
  - Clinique et Maternité Sainte Elisabeth, Namur
  - AZ Damiaan, Ostend
- France (20):
  - Institut Bergonie, Bordeaux
  - CHU de Brest, Brest
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - Centre Hospitalier de la Dracénie, Draguignan
  - CHU de Grenoble - La Tronche - Hôpital A. Michallon, Grenoble
  - Centre Hospitalier Departemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier de Versailles - Hopital Andre Mignot, Le Chesnay
  - CHU de Limoges - Hopital Dupuytren, Limoges
  - Clinique de la Sauvegarde, Lyon
  - Centre Hospitalier D'Annecy, Metz-Tessy
  - Centre Hospitalier de Mont-de-Marsan, Mont-de-Marsan
  - Centre Catherine De Sienne, Nantes
  - Institut Curie, Paris
  - Institut Curie - Hopital Rene Huguenin, Saint-Cloud
  - Hopitaux Universitaires de Strasbourg - Hôpitaux Universitaires de Strasbourg - Hôpital civil, Strasbourg
  - Hopitaux du Leman - Site Georges Pianta, Thonon-les-Bains
  - CH de Valence, Valence
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (50):
  - Klinikum St. Marien, Amberg
  - Gemeinschaftspraxis Augsburg, Augsburg
  - Klinikum Augsburg, Augsburg
  - Praxisklinik Krebsheilkunde für Frauen, Berlin
  - Medizinischen Zentrum Bonn, Bonn
  - Marienhospital Bottrop gGmbH, Bottrop
  - Klinikum Sindelfingen-Boeblingen, Böblingen
  - Gemeinschaftspraxis Lorenz / Hecker / Wesche, Braunschweig
  - Onkologische-Hämatologischen Schwerpunktpraxis, Bremen
  - Universitaetsklinikum Koeln, Cologne
  - Onkologische Gemeinschaftspraxis, Dresden
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Luisenkrankenhaus GmbH & Co. KG, Düsseldorf
  - Universitaetsklinik Duesseldorf, Düsseldorf
  - Universitaetsklinik Erlangen, Erlangen
  - Universitaetsklinikum - Essen, Essen
  - Staedtische Kliniken, Esslingen am Neckar
  - Ev.-Luth. Diakonissenanstalt Flensburg, Flensburg
  - Staedtische Kliniken Frankfurt Am Main-Hoechst, Frankfurt am Main
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaets-Krankenhaus Eppendorf, Hamburg
  - Gynäkologisch-Onkologischen Schwerpunktpraxis, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Gemeinschaftspraxis Dr. Pourfard / Dr. Uleer, Hildesheim
  - St. Marien-Klinik GmbH Frauenklinik der St. Vincentius-Kliniken gAG, Karlsruhe
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Klinikum Landshut, Landshut
  - Staedtisches Klinikum Leipzig - Klinikum St. Georg gGmbH, Leipzig
  - Klinikum Ludwigsburg, Ludwigsburg
  - Gemeinschaftspraxis Dr. Goldmann/ Dr. Ebert, Lüneburg
  - UniversitaetsMedizin Mannheim, Mannheim
  - Klinikum Schwaebisch-Gmuend, Mutlangen
  - Gemeinschaftspraxis Prof. Salat / Dr. Stötzer, München
  - Ludwig-Maximilians-Universitaet Muenchen - Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe - Innenstadt, München
  - Muencher Onkol. Praxis Elisenhof, München
  - Onkologische Praxis Oldenburg, Oldenburg
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - RoMed Klinikum Rosenheim, Rosenheim
  - HELIOS Kliniken - HELIOS Klinik Rottweil, Rottweil
  - HELIOS Kliniken - HELIOS Brustzentrums Nordachsen - HELIOS Klinik Schkeuditz, Schkeuditz
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall
  - Leopoldina-Krankenhaus der Stadt Schweinfurt gGmbH, Schweinfurt
  - Kliniken Landkreis Sigmaringen GmbH, Sigmaringen
  - Klinikum Stuttgart, Stuttgart
  - Klinikum Traunstein, Traunstein
  - Gesellschaft für onkologische Studien, Praxismanagement und -Logistik, Troisdorf
  - Eberhard Karls Universitaet Tuebingen - Universitaetsfrauenklinik Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - Gesundheitszentren Rhein-Neckar - GRN-Klinik Weinheim, Weinheim
  - Onkologische Schwerpunktpraxis Wupperta, Wuppertal
- Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Ignatiadis M, Rack B, Rothe F, Riethdorf S, Decraene C, Bonnefoi H, Dittrich C, Messina C, Beauvois M, Trapp E, Goulioti T, Tryfonidis K, Pantel K, Repollet M, Janni W, Piccart M, Sotiriou C, Litiere S, Pierga JY. Liquid biopsy-based clinical research in early breast cancer: The EORTC 90091-10093 Treat CTC trial. Eur J Cancer. 2016 Aug;63:97-104. doi: 10.1016/j.ejca.2016.04.024. Epub 2016 Jun 10. PMID 27289552
- See also: Related Info — http://www.eortc.be/clinicaltrials/details.asp?protocol=90091